CLINICAL TRIAL: NCT01097031
Title: Continuous or Intermittent for Keeping Arterial Catheter in Children: A Randomized Clinical Trial
Acronym: UP4061
Status: Completed | Type: Observational
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Maria Carolina Witkowski, Instituto de Cardiologia do Rio Grande do Sul
Other Study IDs: UP4061
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Blood Pressure
Keywords: blood pressure; pediatric; nursing; maintenance arterial catheter

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Continuous Infusion
- Intermittent Infusion
- Infusion Continuous
  Interventions: Other: Infusion Intermittent

INTERVENTIONS:
Other: Infusion Intermittent
  Groups: Infusion Continuous

SUMMARY:
Randomized Clinical Trial to evaluate which is the best infusion system of heparin solution for Keeping the mean invasive blood pressure whether the continuous system and the intermittent one.

ELIGIBILITY:
Inclusion Criteria:

* patients in post-operative in congenital heart disease under 15 kg

Exclusion Criteria:

* no consent of parents or responses

Max Age: 93 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with congenital heart disease
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-10; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
blooding | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Witkowski MC, Moraes MA, Firpo CM. Lack of difference between continuous versus intermittent heparin infusion on maintenance of intra-arterial catheter in postoperative pediatric surgery: a randomized controlled study. Rev Paul Pediatr. 2013 Dec;31(4):516-22. doi: 10.1590/S0103-05822013000400015. PMID 24473958